CLINICAL TRIAL: NCT06107036
Title: Thorough QT Study to Evaluate the Effects of BI 1015550 as Single Doses Following Oral Administration on Cardiac Safety Parameters (Double-blind, Randomized, Placebo-controlled, Five-period Crossover, With Open-label Moxifloxacin as Positive Control) in Healthy Male and Female Subjects
Brief Title: A Study in Healthy People to Test Whether Different Doses of BI 1015550 Have Potential to Induce Heart Rhythm Abnormalities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1305-0026; U1111-1295-4664 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This trial will be performed as a randomized, double-blind, 5-period crossover of BI 1015550 and moxifloxacin. Placebo will be given in two separate periods. There will be 15 treatment sequences based on a Prescott triple Latin square design for 5 treatments and 5 periods.
Who Masked: Participant, Investigator
Masking Description: The administration of BI 1015550 and placebo will be blinded while the administration of moxifloxacin will be carried out open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Sequence 1: H/M/P2/L/P1 (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 2: H/P1/L/P2/M (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 3: H/L/P2/M/P1 (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 4: M/H/L/P1/P2 (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 5: M/P1/L/H/P2 (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 6: M/P2/H/L/P1 (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 7: P1/M/H/P2/L (Experimental): Participants in this study received five treatments ordered as described below. Each treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours. Each treatment was separated by a wash-out period of at least 7 days.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 8: P1/P2/H/M/L (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 9: P1/L/M/H/P2 (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 10: P2/H/P1/M/L (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 11: P2/P1/M/L/H (Experimental): Participants in this study received five treatments ordered as described below. Each treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours. Each treatment was separated by a wash-out period of at least 7 days.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 12: P2/L/M/P1/H (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 13: L/H/P1/P2/M (Experimental): Participants in this study received five treatments in the order described below. Each treatment was administered orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 14: L/M/P2/P1/H (Experimental): Participants in this study received five treatments ordered as described below. Each treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours. Each treatment was separated by a wash-out period of at least 7 days.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo
- Sequence 15: L/P2/P1/H/M (Experimental): Participants in this study received five treatments ordered as described below. Each treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours. Each treatment was separated by a wash-out period of at least 7 days.
  L (low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  H (high-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  M (high-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin as a positive control.
  Interventions: Drug: BI 1015550; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: BI 1015550 — BI 1015550 administered as low (L), and high (H), dose. Oral tablet.
  Other Names: Nerandomilast; JASCAYD®
Drug: Moxifloxacin — Moxifloxacin was used as positive control, given as a high dose. Oral tablet.
  Other Names: Avelox®
Drug: Placebo — Placebo was administered as low (P1), matching the low-dose nerandomilast group, and as high (P2), matching the high-dose neradnomilast group. Oral tablet.

SUMMARY:
The main objective of this trial is to evaluate the effects of a single therapeutic and a single supra-therapeutic dose of BI 1015550 following oral administration on cardiac safety parameters in healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs - blood pressure (BP) and pulse rate (PR), 12-lead electrocardiogram (ECG), and clinical laboratory tests without any clinically significant abnormalities
2. Age of 18 to 50 years (inclusive)
3. Body mass index of 18.5 to 32 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. Either male subjects, or female subjects meet the following criteria requiring highly effective contraception from at least 30 days before the first administration of trial medication until 37 days after the last administration of the study drug:

   * Male participants must use condom plus their partner, if identified as a women of childbearing potential (WOCBP), must use an oral contraceptive or highly effective contraception
   * Female participants must be using highly effective contraception and in addition their male partner must use a condom if they are using an oral contraceptive

Exclusion Criteria:

1. Any finding in the medical examination (including BP, Heart rate (HR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or heart rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (alanine transaminase, aspartate transaminase, total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to depression and suicidal behaviour
8. History of clinically relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, placebo-controlled, double-blind (moxifloxacin: open-label), crossover study had 5 treatment periods separated by ≥7-day washouts.
  Treatments included a low dose nerandomilast [L], a high dose nerandomilast [H], a high dose moxifloxacin (positive control) [M]), and placebo [P1, P2].
  The study assessed nerandomilast's effect on cardiac safety (QT/QTc interval) in healthy female and male participants across 15 sequences, each with 3 participants.
Pre-assignment Details: A total of 46 participants who met all inclusion and no exclusion criteria were enrolled in the study, and all completed the planned observation period per protocol. Participants could withdraw from the trial at any time. Two participants were partially excluded from the analysis: one due to a protocol deviation and the other due to the use of rescue medication.
Period: Treated in period 1
Arm/Group | Sequence 1: H/M/P2/L/P1 | Sequence 2: H/P1/L/P2/M | Sequence 3: H/L/P2/M/P1 | Sequence 4: M/H/L/P1/P2 | Sequence 5: M/P1/L/H/P2 | Sequence 6: M/P2/H/L/P1 | Sequence 7: P1/M/H/P2/L | Sequence 8: P1/P2/H/M/L | Sequence 9: P1/L/M/H/P2 | Sequence 10: P2/H/P1/M/L | Sequence 11: P2/P1/M/L/H | Sequence 12: P2/L/M/P1/H | Sequence 13: L/H/P1/P2/M | Sequence 14: L/M/P2/P1/H | Sequence 15: L/P2/P1/H/M
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treated in period 2
Arm/Group | Sequence 1: H/M/P2/L/P1 | Sequence 2: H/P1/L/P2/M | Sequence 3: H/L/P2/M/P1 | Sequence 4: M/H/L/P1/P2 | Sequence 5: M/P1/L/H/P2 | Sequence 6: M/P2/H/L/P1 | Sequence 7: P1/M/H/P2/L | Sequence 8: P1/P2/H/M/L | Sequence 9: P1/L/M/H/P2 | Sequence 10: P2/H/P1/M/L | Sequence 11: P2/P1/M/L/H | Sequence 12: P2/L/M/P1/H | Sequence 13: L/H/P1/P2/M | Sequence 14: L/M/P2/P1/H | Sequence 15: L/P2/P1/H/M
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 (One participant discontinued due to a positive drug test.) | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treated in period 3
Arm/Group | Sequence 1: H/M/P2/L/P1 | Sequence 2: H/P1/L/P2/M | Sequence 3: H/L/P2/M/P1 | Sequence 4: M/H/L/P1/P2 | Sequence 5: M/P1/L/H/P2 | Sequence 6: M/P2/H/L/P1 | Sequence 7: P1/M/H/P2/L | Sequence 8: P1/P2/H/M/L | Sequence 9: P1/L/M/H/P2 | Sequence 10: P2/H/P1/M/L | Sequence 11: P2/P1/M/L/H | Sequence 12: P2/L/M/P1/H | Sequence 13: L/H/P1/P2/M | Sequence 14: L/M/P2/P1/H | Sequence 15: L/P2/P1/H/M
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treated in period 4
Arm/Group | Sequence 1: H/M/P2/L/P1 | Sequence 2: H/P1/L/P2/M | Sequence 3: H/L/P2/M/P1 | Sequence 4: M/H/L/P1/P2 | Sequence 5: M/P1/L/H/P2 | Sequence 6: M/P2/H/L/P1 | Sequence 7: P1/M/H/P2/L | Sequence 8: P1/P2/H/M/L | Sequence 9: P1/L/M/H/P2 | Sequence 10: P2/H/P1/M/L | Sequence 11: P2/P1/M/L/H | Sequence 12: P2/L/M/P1/H | Sequence 13: L/H/P1/P2/M | Sequence 14: L/M/P2/P1/H | Sequence 15: L/P2/P1/H/M
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treated in period 5
Arm/Group | Sequence 1: H/M/P2/L/P1 | Sequence 2: H/P1/L/P2/M | Sequence 3: H/L/P2/M/P1 | Sequence 4: M/H/L/P1/P2 | Sequence 5: M/P1/L/H/P2 | Sequence 6: M/P2/H/L/P1 | Sequence 7: P1/M/H/P2/L | Sequence 8: P1/P2/H/M/L | Sequence 9: P1/L/M/H/P2 | Sequence 10: P2/H/P1/M/L | Sequence 11: P2/P1/M/L/H | Sequence 12: P2/L/M/P1/H | Sequence 13: L/H/P1/P2/M | Sequence 14: L/M/P2/P1/H | Sequence 15: L/P2/P1/H/M
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
Groups:
- All Participants: In this study, all participants received five treatments, administered in 15 different sequences. Each treatment was given orally with 240 mL of water following an overnight fast of at least 10 hours. A washout period of at least 7 days separated each treatment.
  The treatments were as follows:
  H (High-dose nerandomilast): Participants received film-coated tablets containing a high dose of nerandomilast.
  L (Low-dose nerandomilast): Participants received film-coated tablets containing a low dose of nerandomilast.
  M (High-dose moxifloxacin - Positive Control): Participants received film-coated tablets containing a high dose of moxifloxacin, which served as a positive control.
  P1 (Placebo 1): Participants received placebo tablets designed to match the low-dose nerandomilast group.
  P2 (Placebo 2): Participants received placebo tablets designed to match the high-dose nerandomilast group.
Arm/Group | All Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Mean Difference Between Each Single Dose of Either a Low Dose or a High Dose of Nerandomilast and Placebo in QTcF Changes From Baseline Between 20 Min to 24 Hours After Drug Administration
Description: QT interval corrected for heart rate (using the method of Fridericia, QTcF) changes from baseline, measured between 20 minutes and 24 hours after drug administration, were analyzed using a linear Mixed Model for Repeated Measures (MMRM). Pairwise comparison was used to compare the QTcF changes for each dose of nerandomilast (e.g., low dose, high dose) with the placebo at every time point. Mean treatment differences in the QTcF changes from baseline at each time point were estimated by the differences in the corresponding least-squares means. Two-sided 90% confidence intervals based on the t-distribution were computed for each time point. The MMRM was adjusted for the discrete fixed effects treatment, period, time, the continuous fixed effects period- and participant-baseline, the fixed effect-by-time terms, participant as random effect and time within period as a repeated effect per participant. The covariance structure for the repeated effect time was unstructured.
Time Frame: MMRM included measurements at these time points [hours:minutes] post-drug: 0:20, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 4:30, 5:00, 6:00, 8:00, 12:00, and 24:00. MMRM values at 12:00 (low dose) and 4:30 (high dose) are shown in the table below.
Population: Electrocardiogram set (ECGS): This participant set includes all participants in the treated set who have at least one on-treatment value for at least one electrocardiogram (ECG) endpoint, which is not excluded due to ECG relevant important protocol deviations (iPDs). Such iPDs may be e.g., the use of pro-arrhythmic medications. Only participants with available ECG data were included.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Groups:
- Low-dose nerandomilast: Participants who received film-coated tablets containing a low dose of nerandomilast. The treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours.
- High-dose nerandomilast: Participants received film-coated tablets containing a high dose of nerandomilast.
  The treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours.
Arm/Group | Low-dose nerandomilast | High-dose nerandomilast
Number analyzed (Participants) | 43 | 45
Milliseconds | 3.0 [0.7 to 5.4] | 3.2 [1.2 to 5.2]

2. Secondary Outcome: The Maximum Mean Difference Between Moxifloxacin and Placebo in QTcF Changes From Baseline Between 20 Min to 24 Hours After Drug Administration.
Description: QT interval corrected for heart rate (using the method of Fridericia, QTcF) changes from baseline, measured between 20 minutes and 24 hours after drug administration, were analyzed using a linear Mixed Model for Repeated Measures (MMRM). Pairwise comparison was used to compare the QTcF changes for moxifloxacin with the placebo at every time point. Mean treatment differences in the QTcF changes from baseline at each time point were estimated by the differences in the corresponding least-squares means. Two-sided 90% confidence intervals based on the t-distribution were computed for each time point. The MMRM was adjusted for the discrete fixed effects treatment, period, time, the continuous fixed effects period- and participant-baseline, the fixed effect-by-time terms, participant as random effect and time within period as a repeated effect per participant. The covariance structure for the repeated effect time was unstructured.
Time Frame: MMRM included measurements at these time points [hours:minutes] post-drug: 0:20, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 4:30, 5:00, 6:00, 8:00, 12:00, and 24:00. MMRM values at 3:30 (high dose moxifloxacin) are shown in the table below.
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Groups:
- High-dose moxifloxacin - Positive Control: Participants who received film-coated tablets containing a high dose of moxifloxacin as a positive control. The treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours.
  Moxifloxacin was used as a positive control due to its modest QT-prolonging properties at a high dose level.
Arm/Group | High-dose moxifloxacin - Positive Control
Number analyzed (Participants) | 44
Milliseconds | 14.2 [12.4 to 16.1]

ADVERSE EVENTS:
Time Frame: Adverse Events: up to 7 days following drug administration for placebo 1 and 2, low-dose nerandomilast, and high-dose nerandomilast, and for up to 4 days following administration of high-dose moxifloxacin. All-Cause Mortality: from the first drug administration on Day 1 until the end of the trial, up to a total of 44 days.
Description: Treated set (TS): The treated set includes all participants who were treated with at least one dose of trial drug.
Groups:
- Placebo 1: Participants who received placebo tablets designed to match the low-dose nerandomilast group. The treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours.
- Placebo 2: Participants who received placebo tablets designed to match the high-dose nerandomilast group. The treatment was administered orally with 240 mL of water after an overnight fast of at least 10 hours.
Arm/Group | Placebo 1 | Placebo 2 | Low-dose nerandomilast | High-dose nerandomilast | High-dose moxifloxacin - Positive Control
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46 | 0/45 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46 | 0/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 4/46 | 4/45 | 3/45 | 3/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 1 (N=45) | Placebo 2 (N=46) | Low-dose nerandomilast (N=45) | High-dose nerandomilast (N=45) | High-dose moxifloxacin - Positive Control (N=45)
Headache (Nervous system disorders) | 0 | 4 | 4 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT06107036/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT06107036/SAP_001.pdf